CLINICAL TRIAL: NCT04609696
Title: A 2-Part, Open-Label, Randomized, Single-Dose, 3-Period Crossover, Phase 1, Relative Bioavailability, and Food Effect Study, Comparing Different Formulations of Danicopan in Healthy Adult Subjects
Brief Title: Study of the Metabolism of Danicopan in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN2040-HV-119
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Tablet; Capsule; Danicopan; Bioavailability; Factor D Inhibitor; Food Effect
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Sequence 1 (Experimental): Participants will receive danicopan once each period as a single oral dose under fasted or fed conditions as follows:
  Period 1: Danicopan as the PIC 1 formulation under fed conditions. Period 2: Danicopan as the PIC 1 formulation under fasted conditions. Period 3: Danicopan as a tablet under fed conditions.
  There will be a washout period of at least 5 days between each danicopan dosing.
  Interventions: Drug: Danicopan: Powder-In-Capsule 1; Drug: Danicopan: Tablet
- Part 1: Sequence 2 (Experimental): Participants will receive danicopan once each period as a single oral dose under fasted or fed conditions as follows:
  Period 1: Danicopan as the PIC 1 formulation under fasted conditions. Period 2: Danicopan as a tablet under fed conditions. Period 3: Danicopan as the PIC 1 formulation under fed conditions.
  There will be a washout period of at least 5 days between each danicopan dosing.
  Interventions: Drug: Danicopan: Powder-In-Capsule 1; Drug: Danicopan: Tablet
- Part 1: Sequence 3 (Experimental): Participants will receive danicopan once each period as a single oral dose under fasted or fed conditions as follows:
  Period 1: Danicopan as a tablet under fed conditions. Period 2: Danicopan as the PIC 1 formulation under fed conditions. Period 3: Danicopan as the PIC 1 formulation under fasted conditions.
  There will be a washout period of at least 5 days between each danicopan dosing.
  Interventions: Drug: Danicopan: Powder-In-Capsule 1; Drug: Danicopan: Tablet
- Part 2: Sequence 1 (Experimental): Participants will receive danicopan once each period as a single oral dose under fasted or fed conditions as follows:
  Period 1: Danicopan as the PIC 2 formulation under fed conditions. Period 2: Danicopan as the PIC 2 formulation under fasted conditions. Period 3: Danicopan as a tablet under fed conditions.
  There will be a washout period of at least 5 days between each danicopan dosing.
  Interventions: Drug: Danicopan: Powder-In-Capsule 2; Drug: Danicopan: Tablet
- Part 2: Sequence 2 (Experimental): Participants will receive danicopan once each period as a single oral dose under fasted or fed conditions as follows:
  Period 1: Danicopan as the PIC 2 formulation under fasted conditions. Period 2: Danicopan as a tablet under fed conditions. Period 3: Danicopan as the PIC 2 formulation under fed conditions.
  There will be a washout period of at least 5 days between each danicopan dosing.
  Interventions: Drug: Danicopan: Powder-In-Capsule 2; Drug: Danicopan: Tablet
- Part 2: Sequence 3 (Experimental): Participants will receive danicopan once each period as a single oral dose under fasted or fed conditions as follows:
  Period 1: Danicopan as a tablet under fed conditions. Period 2: Danicopan as the PIC 2 formulation under fed conditions. Period 3: Danicopan as the PIC 2 formulation under fasted conditions.
  There will be a washout period of at least 5 days between each danicopan dosing.
  Interventions: Drug: Danicopan: Powder-In-Capsule 2; Drug: Danicopan: Tablet

INTERVENTIONS:
Drug: Danicopan: Powder-In-Capsule 1 — Danicopan (200 milligrams) will be administered orally on Day 1.
  Other Names: ALXN2040; ACH-0144471 (formerly)
  Arms: Part 1: Sequence 1; Part 1: Sequence 2; Part 1: Sequence 3
Drug: Danicopan: Powder-In-Capsule 2 — Danicopan (200 milligrams) will be administered orally on Day 1.
  Other Names: ALXN2040; ACH-0144471 (formerly)
  Arms: Part 2: Sequence 1; Part 2: Sequence 2; Part 2: Sequence 3
Drug: Danicopan: Tablet — Danicopan (200 milligrams) will be administered orally on Day 1.
  Other Names: ALXN2040; ACH-0144471 (formerly)

SUMMARY:
This is a 2-part open-label, randomized, single-dose, 3-sequence, 3-period crossover, relative bioavailability, and food-effect study comparing different formulations of danicopan in healthy adult participants.

DETAILED DESCRIPTION:
For both parts of this study, on Day 1 of each period, participants will receive a single oral dose of danicopan as either the prototype powder-in-capsule (PIC) formulation (1 or 2) under fed conditions, the prototype PIC formulation (1 or 2) under fasting conditions, or the tablet formulation under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. No clinically significant findings at screening (medical history, clinical laboratory profiles, and electrocardiograms).
2. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at screening.
3. Female participants of childbearing potential must either agree to abstinence or to use, with their male partner, a highly effective method of contraception .
4. Non-sterile male participants must agree to abstinence or use a highly effective method of contraception.

Exclusion Criteria:

1. History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
2. History or presence of drug or alcohol abuse within previous 2 years, current tobacco user, or positive drugs-of-abuse screen or alcohol screen at screening or Day -1 of Period 1.
3. History of meningococcal infection, or a first-degree relative with a history of meningococcal infection.
4. History of procedures that could alter absorption or excretion of orally administered drugs.
5. History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
6. Body temperature ≥ 38.0°Celcius at screening or prior to first dosing or history of febrile illness, or other evidence of infection, within 14 days prior to (first) dosing.
7. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before first dosing, whichever is longer.
8. Donation of whole blood from 3 months prior to first dosing, or of plasma from 30 days before first dosing, receipt of blood products within 6 months prior to first dosing, or receipt of a vaccine within 30 days prior to first dosing.
9. Is a female with a positive pregnancy test or who is lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability Of Danicopan Prototype PIC 1 Formulation And Tablet Formulation | Up to 72 hours postdose
  The relative bioavailability of the PIC 1 formulation versus the tablet formulation will be measured by the ratio of select pharmacokinetic (PK) parameters: maximum observed plasma concentration (Cmax), area under the concentration-time curve from time of administration to the last measurable concentration (AUC0-t), and area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-inf).
AUC0-inf Of Danicopan Prototype PIC 1 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose
AUC0-t Of Danicopan Prototype PIC 1 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose
Cmax Of Danicopan Prototype PIC 1 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose
Time to maximum observed plasma concentration (Tmax) Of Danicopan Prototype PIC 1 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose
Relative Bioavailability Of Danicopan Prototype PIC 2 Formulation And Tablet Formulation | Up to 72 hours postdose
  The relative bioavailability of the PIC 2 formulation versus the tablet formulation will be measured by the ratio of select PK parameters: Cmax, AUC0-t, and AUC0-inf.
AUC0-inf Of Danicopan Prototype PIC 2 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose
AUC0-t Of Danicopan Prototype PIC 2 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose
Cmax Of Danicopan Prototype PIC 2 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose
Tmax Of Danicopan Prototype PIC 2 Formulation Under Both Fed And Fasted Conditions | Up to 72 hours postdose

SECONDARY OUTCOMES:
Number Of Participants Receiving Prototype PIC 1 And Tablet With Treatment-emergent Adverse Events Under Fed Conditions | Day 1 (postdose) through follow-up (10 [+/- 2] days dosing on Day 1)
Number Of Participants Receiving Prototype PIC 1 With Treatment-emergent Adverse Events Under Fasted Conditions | Day 1 (postdose) through follow-up (10 [+/- 2] days dosing on Day 1)
Number Of Participants Receiving Prototype PIC 2 And Tablet With Treatment-emergent Adverse Events Under Fed Conditions | Day 1 (postdose) through follow-up (10 [+/- 2] days dosing on Day 1)
Number Of Participants Receiving Prototype PIC 2 With Treatment-emergent Adverse Events Under Fasted Conditions | Day 1 (postdose) through follow-up (10 [+/- 2] days dosing on Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No